CLINICAL TRIAL: NCT01029769
Title: The Switch Study - Efficacy of Early Antipsychotic Switch Versus Maintenance in Patients With Schizophrenia Poorly Responding to Two Weeks of Antipsychotic Treatment
Brief Title: Efficacy of an Early Antipsychotic Switch in Case of Poor Initial Response to the Treatment of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 01KG0910
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2015-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Amisulpride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- initial olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine or amisulpride
- initial amisulpride (Active Comparator)
  Interventions: Drug: Olanzapine or amisulpride
- early responders (Active Comparator)
  Interventions: Drug: Olanzapine or amisulpride
- early non-responders switched (Active Comparator)
  Interventions: Drug: Olanzapine or amisulpride
- ealy non-responders non-switched (Active Comparator)
  Interventions: Drug: Olanzapine or amisulpride

INTERVENTIONS:
Drug: Olanzapine or amisulpride — Oral olanzapine 5mg to 20mg/d OR oral amisulpride 200mg to 800mg/d; both preferably once daily, both encapsulated for blinding

SUMMARY:
The main aim of the trial is to study whether a change of medication in non-responders to a two-weeks antipsychotic drug trial is more effective than continued treatment with the same antipsychotic. Hypothesis: Non-responders who are switched at 2 weeks to another antipsychotic are more frequently in symptomatic remission at week 8 than non-responders who stay on the same antipsychotic

DETAILED DESCRIPTION:
The patients will be randomised to a double-blind 2 week run in phase with fixed doses of either oral amisulpride 800 mg/day or olanzapine 20mg/day.

Those participants who have not responded to treatment at two weeks (PANSS improvement <25%) will be randomised to a 6 week double blind flexible dose phase:

1. Experimental intervention: switch to the other antipsychotic (oral olanzapine 5-20mg/d or oral amisulpride 200-800 mg/d)
2. Control intervention: continuation with the same drug as in the first 2 weeks in flexible dose ranges as above for another six weeks Those participants who have responded at week 2 (≥25% PANSS reduction) will continue on the same drug in flexible dose ranges as above Total duration of intervention per patient: 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with Diagnostic and Statistical Manual of Mental Disorders 4th Edition Text Revision (DSM-IV TR) diagnosis of schizophrenia, schizophreniform or schizoaffective disorder
* PANSS total score at baseline > 75, at least two PANSS psychosis items ≥ 4, Clinical Global Impression of severity score moderately ill or more (≥4)
* Increase in the level of care (outpatient care to day clinic or inpatient care)

Exclusion Criteria:

* contraindication to study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-12; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Leucht, MD, Principal Investigator — Psychiatrische Klinik und Poliklinik fuer Psychiatrie und Psychotherapie der Technischen Universität München am Klinikum rechts der Isar
Locations (1):
- Psychiatrische Klinik und Poliklinik fuer Psychiatrie und Psychotherapie der Technischen Universitaet Muenchen am Klinikum rechts der Isar, Munich, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment at baseline comprises the periods "initial olanzapine" and "initial amisulpride"; a re-randomisation was performed after 2 weeks of treatment; the patient numbers in the second phase of the trial must not be added to the overall participant number at baseline (other three groups all formed in phase II of the trial); NOTE that the groups "early responders", "early non-responders switched", "early non-responders non-switched" become active only in phase II of the trial, not before!!
Groups:
- Initial Olanzapin; Initial Amisulpride; Early Responders; Early Non-responders Switched; Ealy Non-responders Non-switched: Olanzapine or amisulpride: Oral olanzapine 5mg to 20mg/d OR oral amisulpride 200mg to 800mg/d; both preferably once daily, both encapsulated for blinding
Period: Period 1: Initial 2-week Treatment
Arm/Group | Initial Olanzapin | Initial Amisulpride | Early Responders | Early Non-responders Switched | Ealy Non-responders Non-switched
Started | 163 | 164 | 0 | 0 | 0
Completed | 140 | 145 | 0 | 0 | 0
Not Completed | 23 | 19 | 0 | 0 | 0
Period: Period 2: Extended 6-week Treatment
Arm/Group | Initial Olanzapin | Initial Amisulpride | Early Responders | Early Non-responders Switched | Ealy Non-responders Non-switched
Started | 0 | 0 | 140 | 70 | 72
Completed | 0 | 0 | 104 | 60 | 55
Not Completed | 0 | 0 | 36 | 10 | 17

BASELINE CHARACTERISTICS:
Population: Three hundred and twenty-seven patients were randomized in study phase I.
Groups:
- Period 1: Initital 2-week Treatment - Amisulpride: Baseline assessment of period 1 of all patients randomised to amisulpride flexible 200-800 mg/d double blind treatment
- Period 1: Initital 2-week Treatment - Olanzapine: Baseline assessment of period 1 of all patients randomised to olanzapine flexible 5-20 mg/d double blind treatment
- Total: Total of all reporting groups
Arm/Group | Period 1: Initital 2-week Treatment - Amisulpride | Period 1: Initital 2-week Treatment - Olanzapine | Total
Number analyzed (Participants) | 163 | 164 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.1) | 39.3 (10.9) | 39.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 79 | 154
  Male | 88 | 85 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 163 | 164 | 327
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 75 | 75 | 150
  Romania | 88 | 89 | 177

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Symptomatic Remission at Week 8 Comparing the "Switched" With the "Non Switched" Early Non-responders
Description: Remission is defined as a maximum rating of 3 points (equals a severity rating of "mild") in each of all the following eight items of the PANSS (Kay et al.) rating scale: Delusions (P1), unusual thought content (G9), hallucinatory behavior (P3), conceptual disorganization (P2), mannerisms/posturing (G5), blunted affect (N1), social withdrawal (N4) and lack of spontaneity (N6); if one item is >3 the remission status is "no" (non-remission); all times have a rating from 1 to 7, so the min. rating is 8, the max. rating is 56. Remission is a dichotomous item (yes/no) without a specific min. or max. rating
Time Frame: 8 weeks
Population: please note that all patients, regardless of the medication received, were combined in these groups for the primary endpoint analysis solely depending on whether they have met the criteria for "early non-response" at the end of phase I of the trial; so the statistical analysis does not follow the treatment arms in phase I of the trial (patients received alternatively olanzapine or amisulpride, but both types of treatment appear in one and the same analysis group!)
Measure: Count of Participants; unit: Participants
Groups:
- Early Non-responders Non-switched: Olanzapine or amisulpride: Oral olanzapine 5mg to 20mg/d OR oral amisulpride 200mg to 800mg/d; both preferably once daily, both encapsulated for blinding
Arm/Group | Early Non-responders Switched | Early Non-responders Non-switched
Number analyzed (Participants) | 60 | 55
Participants | 41 | 25
Statistical Analysis 1: Comparison: Early Non-responders Switched vs Early Non-responders Non-switched; Irrespective of the initially assigned antipsychotic treatment in period 1 of the trial (2-week-phase), the patients showing little improvement over the two weeks of treatment in period 1 now switched from the initial treatment in period 2 of the trial (6-week-phase) were grouped together as well as the patients non-switched from their initial treatment; Test type: Other — a logistic regression model with "remission" as the dependent variable and "switch" of treatment (yes/no) and PANSS-total score at visit 3 as independent variables was used. Multiple imputation (based upon 20 imputations, primary analysis), last observation carried forward and completers only analyses were performed; p = 0.01, Regression, Logistic — Multiple imputation was performed separately for the switch and non-switch arms and the imputation model included the PANSS total score from all visits from phase II baseline (visit 2) onwards, remission at visit 7 and phase I arm allocation

2. Secondary Outcome: PANSS Total Score Change
Description: The Positive and Negative Syndrome Scale (Kay SR, Fiszbein A, Opler LA: The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophrenia Bull 1987; 13:261-276) is a 30- item inventory assessing the absence or severity of schizophrenia symptoms across three subscales: positive symptoms (items P1-P7, including hallucinatory behavior, delusions, and conceptual disorganization), negative symptoms (items N1-N7, including blunted affect, social and emotional withdrawal, and lack of spontaneity), and general psychopathology symptoms (items G1-G16, including mannerisms and posturing, unusual thought content, and lack of insight). Each item is scored on a scale ranging from 1 (absent) to 7 (extreme), with item ratings incorporating the presence, effects of symptoms on an individuum's thinking, feeling or behaving as well as their severity. The min. sum rating is 30, the max. sum rating is 210.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Non-responders Switched | Ealy Non-responders Non-switched
Number analyzed (Participants) | 60 | 55
units on a scale | -22.8 (19.9) | -17.3 (15.1)

ADVERSE EVENTS:
Time Frame: Entire 8 weeks of treatment
Description: spontaneous reporting
Groups:
- Period 1: Initital 2-week Treatment - Amisulpride Treated Patients: oral amisulpride 200mg to 800mg/d; preferably once daily, encapsulated for blinding
- Period 1: Initital 2-week Treatment - Olanzapine Treated Patients: oral olanzapine 5mg to 20mg/d; preferably once daily, encapsulated for blinding
- Period 2: Extended 6-week Treatment - Early Responders; Period 2: Extended 6-week Treatment - Early Non-responders Not Switched: double blind continuation of treatment as in period 1; oral olanzapine 5mg to 20mg/d; OR oral amisulpride 200mg to 800mg/d; preferably once daily, encapsulated for blinding
- Period 2: Extended 6-week Treatment - Early Non-responders Switched: double blind switch to the alternative drug not used in period 1; oral olanzapine 5mg to 20mg/d; OR oral amisulpride 200mg to 800mg/d; preferably once daily, encapsulated for blinding
Arm/Group | Period 1: Initital 2-week Treatment - Amisulpride Treated Patients | Period 1: Initital 2-week Treatment - Olanzapine Treated Patients | Period 2: Extended 6-week Treatment - Early Responders | Period 2: Extended 6-week Treatment - Early Non-responders Switched | Period 2: Extended 6-week Treatment - Early Non-responders Not Switched
All-Cause Mortality (participants affected / at risk) | 0/163 | 1/164 | 1/140 | 0/70 | 0/72
Serious Adverse Events (participants affected / at risk) | 3/163 | 3/164 | 7/140 | 5/70 | 4/72
Other Adverse Events (participants affected / at risk) | 36/163 | 33/164 | 32/140 | 21/70 | 7/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Initital 2-week Treatment - Amisulpride Treated Patients (N=163) | Period 1: Initital 2-week Treatment - Olanzapine Treated Patients (N=164) | Period 2: Extended 6-week Treatment - Early Responders (N=140) | Period 2: Extended 6-week Treatment - Early Non-responders Switched (N=70) | Period 2: Extended 6-week Treatment - Early Non-responders Not Switched (N=72)
prolongation of hospitalisation (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
hospitalisation (Psychiatric disorders) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 3 (3)
life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
life threatening event (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — suicide attempt
life threatening event (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — lithium intoxication
death (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — acute cholecystitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Initital 2-week Treatment - Amisulpride Treated Patients (N=163) | Period 1: Initital 2-week Treatment - Olanzapine Treated Patients (N=164) | Period 2: Extended 6-week Treatment - Early Responders (N=140) | Period 2: Extended 6-week Treatment - Early Non-responders Switched (N=70) | Period 2: Extended 6-week Treatment - Early Non-responders Not Switched (N=72)
akathisia (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2) | 7 (7) | 3 (3) | 1 (1)
tremor (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7) | 8 (8) | 4 (4) | 2 (2)
weight increase (Metabolism and nutrition disorders) | 7 (7) | 12 (12) | 4 (4) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 4 (4) | 6 (6) | 4 (4) | 1 (1)
Insomnia (Nervous system disorders) | 6 (6) | 8 (8) | 7 (7) | 9 (9) | 2 (2)

LIMITATIONS AND CAVEATS:
Patients with poor response to antipsychotic treatment in the past (treatment resistant patients) were not excluded by definition from study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes